CLINICAL TRIAL: NCT01158820
Title: A Randomized, Placebo-controlled, Concealed Allocation Comparison of Respiratory Depression and Coughing During Bronchoscopy With Dexmedetomidine-ketamine as an Adjunct to Fentanyl-midazolam Sedation
Brief Title: Alternative Sedation During Bronchoscopy
Acronym: DEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 810981
Record Dates: First submitted 2010-06-25; First posted 2010-07-08 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Sedation
Keywords: bronchoscopy
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Midazolam; Fentanyl; Diphenhydramine; Doxylamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): midazolam load fentanyl load midazolam demand fentanyl demand benadryl demand
  Interventions: Drug: Midazolam load; Drug: Fentanyl load; Drug: Midazolam demand; Drug: Fentanyl demand; Drug: Benadryl demand
- dexmedetomidine and ketamine (Active Comparator): dexmedetomidine load ketamine load dexmedetomidine maintenance ketamine maintenance midazolam demand fentanyl demand benadryl demand
  Interventions: Drug: Dexmedetomidine load; Drug: Ketamine load; Drug: Dexmedetomidine maintenance; Drug: Ketamine maintenance; Drug: Midazolam demand; Drug: Fentanyl demand; Drug: Benadryl demand

INTERVENTIONS:
Drug: Dexmedetomidine load — Dexmedetomidine 1 µg/kg prior to bronchoscopy
  Other Names: Precedex; Dexmedetomidine Hydrochloride
  Arms: dexmedetomidine and ketamine
Drug: Ketamine load — Ketamine 30 mg bolus prior to bronchoscopy
  Other Names: Ketalar; Calypsol; Ketamin; Ketaminol; Ketanest; Tekam; Vetalar
  Arms: dexmedetomidine and ketamine
Drug: Midazolam load — 2 mg bolus prior to bronchoscopy
  Other Names: Versed
  Arms: Placebo
Drug: Fentanyl load — 50 µg bolus prior to bronchoscopy
  Other Names: Abstral; Actiq; Fentora; Onsolis
  Arms: Placebo
Drug: Dexmedetomidine maintenance — 0.5 µg/kg/hour for the duration of bronchoscopy (58.5 minutes average)
  Other Names: Precedex; Dexmedetomidine Hydrochloride
  Arms: dexmedetomidine and ketamine
Drug: Ketamine maintenance — 8 µg/kg/min for the duration of bronchoscopy (58.5 minutes average)
  Other Names: Ketalar; Calypsol; Ketamin; Ketaminol; Ketanest; Tekam; Vetalar
  Arms: dexmedetomidine and ketamine
Drug: Midazolam demand — 0.5 mg demand bolus at discretion of pulmonologist
  Other Names: Versed
Drug: Fentanyl demand — 12.5 µg demand bolus at discretion of pulmonologist
  Other Names: Abstral; Actiq; Fentora; Onsolis
Drug: Benadryl demand — 25 mg bolus after 6th and 13th demand midazolam/fentanyl bolus
  Other Names: Diphenhydramine Hcl; Aler-Dryl; Banophen; Ben Tann; Bromanate AF; Diphen; Diphenadryl; Diphenhist; Dytan; Unisom; Sominex; Silphen; Siladryl

SUMMARY:
This protocol hopes to determine whether the use of dexmedetomidine-ketamine can reduce the use of standard of care fentanyl-midazolam sedation during bronchoscopy. This may result in less respiratory depression while providing better compliance with the procedure.

DETAILED DESCRIPTION:
All patients enrolled in the study will be undergoing bronchoscopy, which is typically performed with sedation. All procedural sedation carries some risk. Several features of the study may lower the risk of sedation relative to that of conventional sedation. An anesthesiologist will be present throughout the procedure. Continuous monitoring of respiration with RIP will be employed. Administration of sedation will be via a volumetric syringe pump. Benefits specific to dexmedetomidine-ketamine include the lack of respiratory depression and greater hemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 scheduled for elective flexible bronchoscopy in the endoscopy suite or OR of HUP

Exclusion Criteria:

* History of inability to complete bronchoscopy attributable to inadequate sedation
* Requiring more than 2 LPM supplemental oxygen to maintain SaO2 > 90%
* History of allergy to study medications
* Pregnancy
* A history of psychosis
* Any condition deemed likely by the pulmonologist or anesthesiologist to pose a significant risk due to elevation of blood pressure, including cerebral/aortic aneurysm, and or ischemic cardiovascular disease
* Bradydysrhythmia deemed significant by the anesthesiologist or pulmonologist
* A diagnosis of significant renal or hepatic impairment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff E Mandel, MD MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Yarmus LB, Akulian JA, Gilbert C, Mathai SC, Sathiyamoorthy S, Sahetya S, Harris K, Gillespie C, Haas A, Feller-Kopman D, Sterman D, Lee HJ. Comparison of moderate versus deep sedation for endobronchial ultrasound transbronchial needle aspiration. Ann Am Thorac Soc. 2013 Apr;10(2):121-6. doi: 10.1513/AnnalsATS.201209-074OC. PMID 23607840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the practices of the pulmonologist sub investigators by the principal investigator
Groups:
- Placebo: 1. Nebulized lidocaine 2% (maximum dose 200 mg) will be administered for 20 minutes.
  2. Following nebulization, syringe A (placebo) will be given at a rate of 1 µg/kg (based on a concentration of 4 µg/ml) for 10 minutes. Supplemental topical anesthesia will be administered by the pulmonologist during this time.
  3. After step 2, syringe B (midazolam 2 mg and fentanyl 50 µg) will be administered by the anesthesiologist. The infusion rate of syringe A (placebo) will be decreased to 0.7 µg/kg/hr. Syringe C (placebo) will be infused at 4 µg/kg/min (based on 10 mg/ml concentration)
  4. Boluses of 0.5 mg midazolam and 12.5 µg fentanyl will be administered by the pulmonologist from syringe D as needed for patient comfort. Syringe E (benadryl 25 mg) will be administered in entirety by the anesthesiologist after the 6th and 16th bolus of midazolam/fentanyl.
  placebo + Standard of Care of midazolam and fentanyl: Control Saline 50 ml Midazolam 2 mg + Fentanyl 50 µg Saline 20 ml Midazolam 1
- Dexmedetomidine and Ketamine: 1. Nebulized lidocaine 2% (maximum dose 200 mg) will be administered for 20 minutes.
  2. Following nebulization, syringe A (dexmedetomidine) will be given at a rate of 1 µg/kg (based on a concentration of 4 µg/ml) for 10 minutes. Supplemental topical anesthesia will be administered by the pulmonologist during this time.
  3. After step 2, syringe B (ketamine 30 mg) will be administered by the anesthesiologist. The infusion rate of syringe A (dexmedetomidine) will be decreased to 0.7 µg/kg/hr. Syringe C (ketamine) will be infused at 4 µg/kg/min (based on 10 mg/ml concentration)
  4. Boluses of 0.5 mg midazolam and 12.5 µg fentanyl will be administered by the pulmonologist from syringe D as needed for patient comfort. Syringe E (benadryl 25 mg) will be administered in entirety by the anesthesiologist after the 6th and 16th bolus of midazolam/fentanyl.
  dexmedetomidine and ketamine Study Medication: Experimental Dexmedetomidine 200 µg in 50 ml Ketamine 30 mg Ketamine 200 mg in 20 ml M
Period: Overall Study
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo + Standard of Care of midazolam and fentanyl
- Dexmedetomidine and Ketamine: dexmedetomidine and ketamine + Standard of Care of midazolam and fentanyl
- Total: Total of all reporting groups
Arm/Group | Placebo | Dexmedetomidine and Ketamine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (13.2) | 61.2 (14.9) | 59.88 (15.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 12 | 19 | 31
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Decreased Minute Ventilation
Description: An initial baseline minute ventilation estimate was obtained via calibrated respiratory impedance plethysmography bands. Subsequent minute ventilation was normalized to this value. Values exceeding 100% were excluded from analysis, as these typically reflected a period of hyperpnea subsequent to relief of airway obstruction by chin lift or jaw thrust.
Time Frame: During the bronchoscopy procedure only, 58.5 minutes average
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Groups:
- Dexmedetomidine and Ketamine: dexmedetomidine and ketamine + Standard of Care (Midazolam + fentanyl)
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Number analyzed (Participants) | 25 | 25
percentage of baseline | 0.736 [0.592 to 0.848] | 0.764 [0.592 to 0.891]
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine and Ketamine; Test type: Other — No data available for power analysis; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.028

2. Primary Outcome: Total Fentanyl
Description: Total fentanyl dose delivered during the procedure
Time Frame: During the bronchoscopy procedure only, 58.5 minutes average
Measure: Median (Inter-Quartile Range); unit: µg
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Number analyzed (Participants) | 25 | 25
µg | 112.5 [87.5 to 188.4] | 68.75 [21.9 to 103.1]
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine and Ketamine; See reference power analysis; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 43.75 — units are µg

3. Primary Outcome: Total Midazolam
Description: Total midazolam delivered during procedure
Time Frame: Duration of procedure
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Number analyzed (Participants) | 25 | 25
mg | 4.5 [3.5 to 7.5] | 2.75 [0.9 to 4.1]
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine and Ketamine; See reference for power analysis; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.75 — units are mg

4. Secondary Outcome: Desaturation (Cumulative)
Description: Cumulative time below saturation of 90% - the total number of seconds that the pulse oximeter reported a saturation below 90%
Time Frame: During the bronchoscopy procedure only, 58.5 minutes average
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Number analyzed (Participants) | 25 | 25
seconds | 39 [8.5 to 117.5] | 40 [3.8 to 170.5]

5. Secondary Outcome: Desaturation (Longest)
Description: Longest time below saturation of 90% (the number of seconds elapsed between the start of a period in which the pulse oximeter saturation fell below 90% and the return above 90%)
Time Frame: During the bronchoscopy procedure only, 58.5 minutes average
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Number analyzed (Participants) | 25 | 25
seconds | 21 [5 to 43.5] | 18 [3 to 53.3]

6. Secondary Outcome: Conversion to General Anesthesia
Description: Patients in which the procedure could not be completed without conversion to general anesthesia
Time Frame: During the bronchoscopy procedure only, 58.5 minutes average
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Number analyzed (Participants) | 25 | 25
Participants | 6 | 1

7. Secondary Outcome: Patient Satisfaction
Description: Satisfaction rated by 10 point Likert scale (0 = Totally dissatisfied, 10 = Totally satisfied)
Time Frame: After the bronchoscopy procedure only
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Number analyzed (Participants) | 25 | 25
score on a scale | 9 [7 to 10] | 10 [5 to 10]

8. Secondary Outcome: Endoscopist Satisfaction
Description: Satisfaction rated by 10 point Likert scale (0 = Totally dissatisfied, 10 = Totally satisfied)
Time Frame: After the bronchoscopy procedure only
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Dexmedetomidine and Ketamine
Number analyzed (Participants) | 25 | 25
score on a scale | 7 [5.5 to 8.5] | 8 [6 to 9.5]

ADVERSE EVENTS:
Time Frame: The AE data was collected over a 2 year period from the enrollment date for each participant .
Groups:
- Placebo: Placebo + Standard of Care (midazolam and fentanyl)
Arm/Group | Placebo | Dexmedetomidine and Ketamine
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
The presence of an anesthesiologist may have affected the aggressiveness of the pulmonologists in administering sedation.

Alterations in the study drug were not permitted; an open label study might find larger differences in respiratory measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes